CLINICAL TRIAL: NCT02715050
Title: Phototherapy Applied in Association With Muscular Training: Evaluation of Different Moments of Applications
Brief Title: Phototherapy Applied in Association With Muscular Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Adriane Aver Vanin, Phd researcher, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PhD437.894
Record Dates: First submitted 2016-03-11; First posted 2016-03-22 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Muscle Adaptation
Keywords: phototherapy; photobiostimulation; muscle training; muscular adaptation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A - Active or Placebo Phototherapy (Experimental): Participants enrolled in this group performed a training protocol for 12 weeks with light application before and after the exercise protocol. The phototherapy device was divided in program 1 and program 2. One of these programs consisted in active phototherapy and the other placebo.
  The subjects allocated in group A, received program 1 before strength training, and the same program 1 after training.
  Interventions: Device: Active or Placebo Phototherapy (MR4)
- Group B - Active or Placebo Phototherapy (Experimental): Participants enrolled in this group performed a training protocol for 12 weeks with light application before and after the exercise protocol. The phototherapy device was divided in program 1 and program 2. One of these programs consisted in active phototherapy and the other placebo.
  The subjects allocated in group B, received program 1 before strength training, and program 2 after training.
  Interventions: Device: Active or Placebo Phototherapy (MR4)
- Group C - Active or Placebo Phototherapy (Experimental): Participants enrolled in this group performed a training protocol for 12 weeks with light application before and after the exercise protocol. The phototherapy device was divided in program 1 and program 2. One of these programs consisted in active phototherapy and the other placebo.
  The subjects allocated in group C, received program 2 before strength training, and program 1 after training.
  Interventions: Device: Active or Placebo Phototherapy (MR4)
- Group D - Active or Placebo Phototherapy (Experimental): Participants enrolled in this group performed a training protocol for 12 weeks with light application before and after the exercise protocol. The phototherapy device was divided in program 1 and program 2. One of these programs consisted in active phototherapy and the other placebo.
  The subjects allocated in group D, received program 2 before strength training, and program 2 after training.
  Interventions: Device: Active or Placebo Phototherapy (MR4)

INTERVENTIONS:
Device: Active or Placebo Phototherapy (MR4)
  Other Names: MR4 device - device that combines super-pulsed lasers, and red and infrared LEDs (Multi Radiance Medical, Solon, OH, USA)

SUMMARY:
The effects of phototherapy has been widely studied by some research groups. The investigators know that there are positive results with light application to improve muscle performance and delay fatigue. However, there are few studies showing its´ effects on muscular training. Therefore, the aim of this study was to assess the effects of phototherapy applied at different times during 12 weeks of strength training. For such, 48 volunteers, healthy male, from 18 to 35 years old were recruited to perform a strength training protocol for the anterior muscle of the thigh development. Volunteers performed the training protocol three times a week for 12 weeks. There were assessed isometric peak torque in isokinetic dynamometer, concentric peak torque, 1-repetition maximum test in the leg extension and leg press machines and bilateral thigh perimetry.

DETAILED DESCRIPTION:
This is a clinical, randomized, controlled placebo and double-blind study. Forty-eight participants performed muscular training protocol. Subjects practiced a protocol training with 60% of the load followed by 80% of the load, measured through 1-repetition maximum test, in all sessions of the training protocol. The training protocol consisted in performing 3 sets of 7 repetitions with 60% of 1-RM, and 4 set of 7 repetitions with 80% of 1-RM. This protocol was performed in every sessions, three times a week, employing leg press and leg extension machines.

Phototherapy, active or placebo, were applied in 6 different points of anterior muscle of the thigh before and after each training session. Only one investigator, that did not participate in any phase of the assessments and trainings sessions, knew about what program is active or placebo in phototherapy device. Randomisation carried out by a simple drawing of lots (A, B, C, or D) in the first visit. The phototherapy unit emitted the same sound regardless of the program used, active or placebo. Either strength training lasted 12 weeks and assessments were performed at baseline, 4, 8 and 12 weeks. There were evaluated maximal voluntary contraction (MVC), concentric torque, bilateral thigh perimetry and 1-repetition maximum test (1-RM).

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals,
* active, that performed less than two exercise sessions per week
* when they presented musculoskeletal injury to the hips or knees in the previous 2 months,
* used pharmacological agents or nutritional supplements regularly, and
* Subjects that did not attend a minimum rate of 80% of all strength training sessions
* Suffered musculoskeletal injury during the ongoing of the study were also excluded.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline Maximum voluntary contraction in the isokinetic dynamometer (MVC) at 12 weeks | 12 weeks
  Functional performance measure - performed in baseline, 4 weeks, 8 weeks and 12 weeks after the beginning of the muscular training
Change from baseline Concentric Torque at 12 weeks | 12 weeks
  Functional performance measure - performed in baseline, 4 weeks, 8 weeks and 12 weeks after the beginning of the muscular training

SECONDARY OUTCOMES:
1-RM test | 12 weeks
  Functional performance measure - performed in baseline, 4 weeks, 8 weeks and 12 weeks after the beginning of the muscular training. This test estimated the load of the exercises.

OTHER OUTCOMES:
Thigh perimetry | 12 weeks
  Muscle mass measure - performed in baseline, 4 weeks, 8 weeks and 12 weeks after the beginning of the muscular training.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Leal-Junior, PhD, Study Director — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Leal-Junior EC, Vanin AA, Miranda EF, de Carvalho Pde T, Dal Corso S, Bjordal JM. Effect of phototherapy (low-level laser therapy and light-emitting diode therapy) on exercise performance and markers of exercise recovery: a systematic review with meta-analysis. Lasers Med Sci. 2015 Feb;30(2):925-39. doi: 10.1007/s10103-013-1465-4. Epub 2013 Nov 19. PMID 24249354
- [Background] Seynnes OR, de Boer M, Narici MV. Early skeletal muscle hypertrophy and architectural changes in response to high-intensity resistance training. J Appl Physiol (1985). 2007 Jan;102(1):368-73. doi: 10.1152/japplphysiol.00789.2006. Epub 2006 Oct 19. PMID 17053104
- [Result] Antonialli FC, De Marchi T, Tomazoni SS, Vanin AA, dos Santos Grandinetti V, de Paiva PR, Pinto HD, Miranda EF, de Tarso Camillo de Carvalho P, Leal-Junior EC. Phototherapy in skeletal muscle performance and recovery after exercise: effect of combination of super-pulsed laser and light-emitting diodes. Lasers Med Sci. 2014 Nov;29(6):1967-76. doi: 10.1007/s10103-014-1611-7. Epub 2014 Jun 19. PMID 24942380